CLINICAL TRIAL: NCT02507414
Title: Characterization of the Mesenteric Traction Syndrome During Upper Gastrointestinal Surgery for Malignant Disease
Brief Title: Mesenteric Traction Syndrome During Upper Gastrointestinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Rikard Ambrus, MD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-3-2014-021
Record Dates: First submitted 2015-07-13; First posted 2015-07-24 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Gastrointestinal Neoplasms; Mesenteric Traction Syndrome
Keywords: Mesenteric Traction Syndrome; Upper gastrointestinal cancer surgery
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Blood Specimen Collection; Head-Down Tilt

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group 1 (Experimental): Patients under going Whipple's procedure, gastric resection and liver resection (n=75).
  Interventions:
  Blood samples obtained pre-, intra-, and one day postoperatively (n=15).
  Measurements of microcirculation using LSCI from procedure start and up to 60 min during surgery.
  Head down tilt of 20 degrees at three time points.
  Interventions: Other: Blood samples; Other: Measurement of microcirculation; Other: Head down tilt

INTERVENTIONS:
Other: Blood samples — 15 arterial blood samples (pre-, intra- and one day postoperatively); no more than 180ml in total over two days.
Other: Measurement of microcirculation — Measurement of microcirculation with Laser Speckle Contrast Imaging (non-touch setup with no side effects); continuous measurement of the microvascular blood flow on the forehead up to 60 minutes starting one minute before the surgical procedure.
  Other Names: LSCI
Other: Head down tilt — At three different time points the participants will be head down tilted in 20 degrees.
  End of surgery (A) One hour postoperatively (B) 18 hours postoperatively (C)

SUMMARY:
It is the hypothesis of this project that the Mesenteric Traction Syndrome (MTS) is a common event during upper gastrointestinal cancer surgery (UGC surgery) and that the induction of the syndrome is an important factor in provoking further peri- and postoperative complications and in worsening the surgical stress response (SSR). The characteristics of MTS is hypotension, tachycardia, and flushing.

In order to uncover the role of MTS in cancer surgery and the effects on the oncological patients, the aim of the project is:

1. To characterize MTS in patients undergoing three common forms of UGC surgery using a new objective methodology and by recording biomarkers suspected of playing a role in the pathophysiology of MTS and postoperative complication development.

Three different interventions will be examined during this prospective trial:

1. Continuous measurement of microcirculation on the forehead using Laser Speckle Contrast Imaging during surgery.
2. Analyses of plasma samples obtained pre-, intra-, and one day postoperatively.
3. Continuous measurements of haemodynamic variables during surgery.

DETAILED DESCRIPTION:
Background

Surgical procedures for upper gastrointestinal cancer (UGC) induce a considerable risk of morbidity and mortality, and more than half of all UGC patients die within one year of diagnosis. Radical surgery is crucial to survival, but is associated with a high risk of complications which contributes to a poor long-term prognosis. Despite advances in surgical techniques and perioperative management, postoperative complications frequently occur.

An essential part of gastrointestinal cancer surgery is the reconstruction of the digestive tract by forming a gut-to-gut reconnection, an anastomosis. Especially during UGC surgery this reconstructive anastomosis is at high risk of insufficient healing and can thus leak intestinal contents into the surrounding tissues, causing life-threatening infections. Development of measures that can reduce the perioperative complications in these vulnerable patients is therefore of vital importance

Patients undergoing surgery for UGC are subjected to a substantial trauma reaction termed the surgical stress response (SSR). SSR is characterized by activation of the sympathetic nervous system, the endocrine system, as well as by immunological and hematological responses leading to hypotension, systemic and local inflammation. In addition, surgical stress can cause immunosuppression in response to the complex interaction of various hormones, cytokines and acute phase reactants. Furthermore, it has recently been reported that perioperative immunosuppression increases the incidence of cancer recurrence, growth of metastases and reduces survival.

A contributing factor to SSR, and possibly most importantly, to the rate of postoperative complications, may be the mesenteric traction syndrome (MTS). MTS arises when the organs of the abdomen are manipulated during surgery. One of the main symptoms is substantial circulatory changes (hypotension, tachycardia and subsequent flushing), which can potentially lead to surgical complications.

Hypothesis and aim

It is the hypothesis of this project that the Mesenteric Traction Syndrome (MTS) is a common event during UGC-surgery and that the induction of the syndrome is an important factor in provoking further peri- and postoperative complications and in worsening the SSR. In order to uncover the role of MTS in cancer surgery and the effects on the oncological patients, the aim of the project is:

To characterize MTS in patients undergoing three common forms of UGC surgery using a new objective methodology and by recording biomarkers suspected of playing a role in the pathophysiology of MTS and postoperative development of complications.

Methods

75 patients undergoing UGC surgery (25 each of the three most common cancer types of UGC) will be included. This study will use a novel skin flushing measuring method called laser speckle contrast imaging (LSCI) to measure skin blood flow of the forehead. LSCI is a real-time and non-touch measuring device capable of measuring blood flow on a large field surface (15 cm x 20 cm). In parallel, inflammatory and hormonal stress biomarkers considered to be associated with SSR, will be measured. In this study, it is hypothesized, that by correlating a new method of quantifiable flushing measurement and known biomarkers, it is possible to relate the extent of flushing to the severity of hypotension and MTS and by proxy the extent of complications.

Furthermore, the participants will be exposed to head down tilt at three pre defined time points with subsequent monitoring of haemodynamics and SSR. This intervention is done to assess the patients' fluid status in the end of surgery as well as postoperatively, as hypovolemia is associated with postoperative complications.

Statistics

The incidence of MTS in UGC patients was previously unknown and power calculations was performed based on previous reported cases of MTS during abdominal surgery (incidence of 30% and 85%). 15 patients are required in each group in order to obtain a statistical power greater than 0.90 with an α-level of < 0.05,. Groups of 25 patients are therefore chosen to ensure statistical significance.

ELIGIBILITY:
Inclusion Criteria:

- patients under going either whipple's procedure, liver resection, or gastric resection.

Exclusion Criteria:

* Robotic assisted procedures
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Relative changes in plasma-hormone concentrations (pro-ANP, PGF2, GLP-1, ACTH, cortisone, adrenaline, IL-1, IL-6, TNF-alfa and CRP (stress hormones)) from baseline. | 15 blood samples obtained pre-, intra-, and 18 hours postoperatively
  A: the day before the surgical procedure B: After induction of anaesthesia (baseline) C: 5 min intraoperatively D: 15 min intraoperatively E: 30 min intraoperatively F: 60 min intraoperatively G: 90 min intraoperatively H: 120 min intraoperatively I: 180 min intraoperatively J: Procedure ending K: 5 min after head down tilt (1) L: One hour after surgery M: 5 min after head down tilt (2) N: 18 hours postoperatively O: 5 min after head down tilt (3)

SECONDARY OUTCOMES:
Postoperative complications | Participants will be followed during the hospital stay, with an expected average of ten days
  All complications will be registered on every postoperative day until discharge.
Relative changes in heart rate from baseline measured in beats per minute | Continuous measurements intra- and postoperatively.
  The variable will be obtained during the surgical procedure using modelflow (Nexfin, BMEYE B.V. Amsterdam, Holland)
Relative changes in microcirculation from baseline during surgery measured in flux-units | A continuous measurement starting one minute prior to the surgical procedure and terminates after 60 minutes.
  Laser Speckle Contrast Imaging (LSCI) is a real-time and non-touch measuring device capable of measuring blood flow on a large field surface (0.5 cm x 0.7 cm up to 15 cm x 20 cm). The infrared LSCI camera is placed at a distance of 20-30 cm and measures the relative flow (flux) at a depth of 1-2 mm by infrared light reflected from circulating erythrocytes in the micro-vessels. The technique will be used for quantifying facial flushing (i.e. increased blood flow to the facial region) during the first hour of surgery, when the MTS is frequently observed.
30-days and 90-days mortality | 30-days and 90-days mortality
Length of stay | Expected time frame of 10 days in average.
Relative changes in median arterial pressure from baseline measured in mmHg | Continuous measurements intra- and postoperatively.
  The variable will be obtained during the surgical procedure using modelflow (Nexfin, BMEYE B.V. Amsterdam, Holland)
Relative changes in cardiac output from baseline measured in litres per minute | Continuous measurements intra- and postoperatively.
  The variable will be obtained during the surgical procedure using modelflow (Nexfin, BMEYE B.V. Amsterdam, Holland)
Relative changes in systemic vascular resistance from baseline measured in dyn.s/cm5 | Continuous measurements intra- and postoperatively.
  The variable will be obtained during the surgical procedure using modelflow (Nexfin, BMEYE B.V. Amsterdam, Holland)

REFERENCES:
- [Background] Rizk NP, Bach PB, Schrag D, Bains MS, Turnbull AD, Karpeh M, Brennan MF, Rusch VW. The impact of complications on outcomes after resection for esophageal and gastroesophageal junction carcinoma. J Am Coll Surg. 2004 Jan;198(1):42-50. doi: 10.1016/j.jamcollsurg.2003.08.007. PMID 14698310
- [Background] Biere SS, van Berge Henegouwen MI, Maas KW, Bonavina L, Rosman C, Garcia JR, Gisbertz SS, Klinkenbijl JH, Hollmann MW, de Lange ES, Bonjer HJ, van der Peet DL, Cuesta MA. Minimally invasive versus open oesophagectomy for patients with oesophageal cancer: a multicentre, open-label, randomised controlled trial. Lancet. 2012 May 19;379(9829):1887-92. doi: 10.1016/S0140-6736(12)60516-9. Epub 2012 May 1. PMID 22552194
- [Background] Giannoudis PV, Dinopoulos H, Chalidis B, Hall GM. Surgical stress response. Injury. 2006 Dec;37 Suppl 5:S3-9. doi: 10.1016/S0020-1383(07)70005-0. PMID 17338909
- [Background] Kehlet H. The stress response to surgery: release mechanisms and the modifying effect of pain relief. Acta Chir Scand Suppl. 1989;550:22-8. PMID 2652970
- [Background] Pham TH, Perry KA, Enestvedt CK, Gareau D, Dolan JP, Sheppard BC, Jacques SL, Hunter JG. Decreased conduit perfusion measured by spectroscopy is associated with anastomotic complications. Ann Thorac Surg. 2011 Feb;91(2):380-5. doi: 10.1016/j.athoracsur.2010.10.006. PMID 21256274
- [Background] Avgerinos DV, Theoharides TC. Mesenteric traction syndrome or gut in distress. Int J Immunopathol Pharmacol. 2005 Apr-Jun;18(2):195-9. doi: 10.1177/039463200501800202. PMID 15888243
- [Background] Seltzer JL, Ritter DE, Starsnic MA, Marr AT. The hemodynamic response to traction on the abdominal mesentery. Anesthesiology. 1985 Jul;63(1):96-9. doi: 10.1097/00000542-198507000-00015. No abstract available. PMID 4014775
- [Background] Mythen MG, Webb AR. Intra-operative gut mucosal hypoperfusion is associated with increased post-operative complications and cost. Intensive Care Med. 1994;20(2):99-104. doi: 10.1007/BF01707662. PMID 8201106
- [Background] Ceppa EP, Fuh KC, Bulkley GB. Mesenteric hemodynamic response to circulatory shock. Curr Opin Crit Care. 2003 Apr;9(2):127-32. doi: 10.1097/00075198-200304000-00008. PMID 12657975